CLINICAL TRIAL: NCT06108622
Title: Prevelance Of Cutaneous Disorders Among Patients With Heamatologic Malignancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Taha, Resident of dermatology ,venerology and andrology department-sohag hospital of mental health, Sohag University
Other Study IDs: soh-Med-23-10-06MS
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Dermatologic Disorders With Heamatologic Malignancies Patients

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cbc ,u\s renalor hepatic function test if needed — just blood sample if the case needed

SUMMARY:
Hematologic malignancies are a diverse group of neoplasms that can have a wide range of clinical and behavioral characteristics. Infections are also a common complication of hematologic malignancies, and can manifest as cutaneous eruptions. Hair loss is a common symptom of hematological malignancies. Changes in the nails can also occur in patients with hematological malignancies. Chemotherapy and radiotherapy are two common treatments for hematological malignancies. patients may experience a wide range of side effects, including hair loss, changes in the nails, and mucositis (

DETAILED DESCRIPTION:
hematologic malignancies are a diverse group of neoplasms that can have a wide range of clinical and behavioral characteristics. The skin is often involved in these diseases, either through direct infiltration by malignant cells or through non-specific changes such as pallor and ecchymosis. Cutaneous involvement can have a significant impact on the quality of life of patients with hematologic malignancies and can also compromise prognosis in certain cases Cutaneous manifestations of hematologic malignancies have become increasingly common. This is partly due to the availability of new drugs that have improved the prognosis of these patients, but also come with an increased risk of skin toxicity. Furthermore, the effectiveness of these therapies has led to increased survival, which in turn has allowed for the emergence of skin eruptions that were not as frequently seen in the past due to the shorter duration of the natural history of cancer Some of the most common manifestations include petechiae, purpura, erythroderma, palpable purpura, Sweet's syndrome and paraneoplastic pemphigus Infections are also a common complication of hematologic malignancies, and can manifest as cutaneous eruptions. For example, patients with leukemia and other blood cancers are at increased risk for developing fungal infections such as candidiasis and aspergillosis, which can present as red, scaly, and itchy skin. Other infections, such as cellulitis, can also occur as a complication of hematologic malignancies and can present with red, swollen, and warm skin Hair loss is a common symptom of hematological malignancies. The cancer cells can interfere with the growth and maintenance of hair follicles, leading to hair loss. Hair loss can be patchy or diffuse, and can occur on the2 scalp, face, or body. In some cases, hair loss can be 2ry to treatment or sign of the progression of the disease. Changes in the nails can also occur in patients with hematological malignancies. The nails may become discolored, brittle, or develop ridges or grooves. In some cases, the nails may also separate from the nail bed. These changes are typically caused by the cancer cells affecting the blood flow to the nails or by the cancer treatment Mucous membranes can also be affected by hematological malignancies. The cancer cells can cause inflammation, soreness, and dryness in the mucous membranes, leading to a condition called mucositis. Mucositis can make it difficult to eat or speak, and can increase the risk of infection. Chemotherapy and radiotherapy are two common treatments for hematological malignancies. These treatments are designed to kill cancer cells or shrink tumors, but they can also affect healthy cells in the body. As a result, patients may experience a wide range of side effects, including hair loss, changes in the nails, and mucositis

. Other common side effects of chemotherapy include nausea, vomiting, fatigue, and an increased risk of infection. Radiation therapy can cause skin reactions, fatigue, and a risk of secondary cancer. Side effects can vary widely depending on the type of cancer and the specific drugs and radiation regimens used. Each patient may experience different side effects, and the intensity and duration of the side effects also vary

ELIGIBILITY:
Inclusion Criteria:

* Age: all age groups.

  * Sex: both sex will be included.
  * Patients with confirmed diagnosis of haematological malignancies ethier clinically or laboratory.

Exclusion Criteria:

* Pregnancy., • Patients with medical comorbidities (liver ,renal ,thyroid abnormalities ,other malignancies)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * A cross - sectional study will include patients who attending and/or admitted to Clinical Oncology and Nuclear Medicine Department Sohag university Hospital.
  * The study protocol will be approved by the Local Ethics and scientific Committee in Sohag faculty of medicine .
  * Written informed consents will be obtained from all patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Prevelance Of Cutaneous Disordera Amog Patients with Heamatologic Malignancies | 1 year
  - A cross - sectional study will include patients who attending and/or admitted to Clinical Oncology and Nuclear Medicine Department Sohag university Hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Atkins S, He F. Chemotherapy and Beyond: Infections in the Era of Old and New Treatments for Hematologic Malignancies. Infect Dis Clin North Am. 2019 Jun;33(2):289-309. doi: 10.1016/j.idc.2019.01.001. Epub 2019 Mar 30. PMID 30935703
- [Background] Didona D, Fania L, Didona B, Eming R, Hertl M, Di Zenzo G. Paraneoplastic Dermatoses: A Brief General Review and an Extensive Analysis of Paraneoplastic Pemphigus and Paraneoplastic Dermatomyositis. Int J Mol Sci. 2020 Mar 21;21(6):2178. doi: 10.3390/ijms21062178. PMID 32245283
- [Background] Dika E, Patrizi A, Veronesi G, Manuelpillai N, Lambertini M. Malignant cutaneous tumours of the scalp: always remember to examine the head. J Eur Acad Dermatol Venereol. 2020 Oct;34(10):2208-2215. doi: 10.1111/jdv.16330. Epub 2020 Apr 7. PMID 32119157
- [Background] Liu YQ, Wang XL, He DH, Cheng YX. Protection against chemotherapy- and radiotherapy-induced side effects: A review based on the mechanisms and therapeutic opportunities of phytochemicals. Phytomedicine. 2021 Jan;80:153402. doi: 10.1016/j.phymed.2020.153402. Epub 2020 Oct 31. PMID 33203590